CLINICAL TRIAL: NCT04863742
Title: Evaluation Of Vision Recovery And Comfort Index In Patients With Borderline/Mild Dry Eyes Undergoing Femtosecond Laser-Assisted Cataract Surgery With Premium Intraocular Lens - The ENHANCE Study
Brief Title: Evaluation Of Vision Recovery And Comfort Index In Patients With Borderline/Mild Dry Eyes Undergoing FLACS With Premium IOL
Acronym: ENHANCE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sight Medical Doctors PLLC (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. John Passarelli, Principle Investigator, Sight Medical Doctors PLLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENHANCE
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Calcium Dobesilate; prednisolone acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dextenza Arm (Experimental)
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Prednisolone Acetate 1% (Active Comparator)
  Interventions: Drug: Prednisolone Acetate

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — sustained released dexamethasone, 0.4mg
  Arms: Dextenza Arm
Drug: Prednisolone Acetate — Prednisolone Acetate 1% QID x 1week, TID x 1week, BID x1 week, QD x1 week.
  Arms: Prednisolone Acetate 1%

SUMMARY:
This is a prospective, open-label, single-center, randomized, head-to-head, investigator-sponsored clinical study. It aims to investigate the vision recovery and patient comfort in borderline/mild dry eye disease patients undergoing FLACS with Premium PCIOL (i.e., Panoptix, Toric IOL (spherical/multifocal), ReStor, Symfony), receiving a 0.4mg dexamethasone intracanalicular insert when compared to patients receiving standard of care prednisolone acetate 1%.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-center, randomized, head-to-head, investigator-sponsored clinical study. It aims to investigate the vision recovery and patient comfort in borderline/mild dry eye disease patients undergoing FLACS with Premium PCIOL (i.e., Panoptix, Toric IOL (spherical/multifocal), ReStor, Symfony), receiving a 0.4mg dexamethasone intracanalicular insert when compared to patients receiving standard of care prednisolone acetate 1%. After screening a given patient for inclusion and exclusion criteria, and gaining informed consent, a total of 30 patients will be randomized into two groups:

Group 1: 15 patients will undergo bilateral FLACS + Premium PCIOL in separate days and will receive a 0.4mg dexamethasone intracanalicular insert at the days of each surgery.

Group 2: 15 patients will undergo bilateral FLACS + Premium PCIOL in separate days and will receive prednisolone acetate 1% QID/ 1 week, TID/ 1 week, BID/1 week, QD/ 1 week regimen starting at the days of each surgery.

All patient eyes will receive Prolensa 0.07% ophthalmic solution QD for 4 weeks starting 3 days prior to surgery and Besivance 0.6% eye drops TID/starting 3 days prior to surgery.

Per enrolled eye, the study period will last for approximately 30 days after surgery, consisting of three postop follow-up visits (six total postop visits per patient). At Day 1, Day 7 and Day 30, primary and secondary endpoints will be assessed alongside standard-of-care procedures. SPEED questionnaire will be assessed by a masked survey administrator. Adjusting for enrollment period, the study will last a total of approximately 12 months, including submission for publication/ presentation.

ELIGIBILITY:
Inclusion Criteria:

1. Demonstrate objective signs of Boderline/ Mild Ocular Surface Disease (OSD) [defined as mild symptoms, mild conjunctival staining (<2+ Superficial Punctate Keratitis), Tear Break-up Time <12s] or demonstrate symptoms of OSD determined by SPEED questionnaire (SPEED Score <10).
2. Nucleus sclerosis up to 2+ planning to undergo FLACS + Premium PCIOL in both eyes.
3. Ability to provide informed consent for procedures
4. Ability to attend scheduled follow up visits
5. No other corneal pathology to create unknown variability

Exclusion Criteria:

1. Age less than 18
2. Pregnancy/currently breast-feeding
3. Inability to provide informed consent
4. Documented adverse reaction to steroid (e.g. "steroid responder", allergy, etc)
5. Punctal stenosis
6. Previous corneal transplant surgery or refractive surgery
7. Concurrent use of topical steroid eye drops
8. Systemic, topical or intravitreal steroid use within 1 month of baseline
9. Active history of chronic or recurrent inflammatory eye disease in either eye
10. History of ocular herpetic infection (inclusive of Herpes Simplex 1/2, Varicella Zoster, Epstein Barr, Cytomegalovirus)
11. History of neurotrophic keratitis, uncontrolled diabetes, or other disease entities that may preclude proper healing
12. Diagnosis of Glaucoma or use of topical glaucoma drops
13. Participation in other studies in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-26 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) | Baseline, Post-Operative Day 7 and Day 30
  As measured by Best Corrected Visual Acuity (BCVA) from baseline and at 1 week and 30 days after surgery
Mean change in uncorrected Visual Acuity (VA) | Baseline, Post-Operative Day 7 and Day 30
  As measured by uncorrected VA from baseline and at 1 week and 30 days after surgery
Mean change from baseline in Standardized Patient Evaluation of Eye Dryness (SPEED) score | Baseline, Post-Operative Day 7 and Day 30
  As measured by SPEED score from baseline and at 1 week and 30 days after surgery

SECONDARY OUTCOMES:
Patient satisfaction with vision at 1 week and 30 days after surgery | Post-Operative Day 7 and Day 30
  As measured by patient satisfaction survey
Mean number of artificial tear drops dosed per day | 30 Day tear log.
  As measured by patient daily log.
Mean change in tear break-up time (TBUT) | Baseline and at POD 7 and POD 30
  As measured by TBUT
Mean change in tear osmolarity | Baseline and at POD 7 and POD 30
  As measured by tear osmolarity
Mean change in corneal staining | Baseline and at POD 7 and POD 30
  As measured by corneal staining
Mean change from baseline in (Central Subfield Thickness) CST | Post-Operative Day 7 and 30
  As measured by CST

CONTACTS AND LOCATIONS:
Overall Officials: John Passarelli, MD, Principal Investigator — Sight Medical Doctors PLLC
Locations (1):
- SightMD, LIASC, Brentwood, New York, United States